CLINICAL TRIAL: NCT07029412
Title: A Phase 2a, Open-label, Exploratory Study to Evaluate Preliminary Efficacy of Subcutaneous MBX 1416 in Patients With Postbariatric Hypoglycemia (The STEADI Study)
Brief Title: Study to Evaluate Efficacy and Dose Response of Imapextide (STEADI)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: MBX Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MBX-1P2002
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Postbariatric Hypoglycemia
Keywords: PBH

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MBX 1416 (INN imapextide) (Experimental): Single subcutaneous administration at different dose levels
  Interventions: Drug: MBX 1416 (INN imapextide)

INTERVENTIONS:
Drug: MBX 1416 (INN imapextide) — A single subcutaneous injection of MBX 1416 at a low dose and a high dose approximately 2 weeks apart.

SUMMARY:
The purpose of this study is to assess the preliminary efficacy of single SC administration of MBX 1416 at different dose levels in patients with PBH

DETAILED DESCRIPTION:
This is a Phase 2a, open-label, exploratory study to evaluate preliminary efficacy of SC MBX 1416 in patients with PBH. Approximately 10 patients aged 18 to 75 (inclusive) years with history of hypoglycemia following Roux-en-Y or sleeve gastrectomy will be included in the study. Participants will undergo 3 mixed-meal tolerance tests, one at baseline and again 48 hours after each MBX 1416 administration, to evaluate the effect of MBX 1416 on increasing post-prandial glucose nadir. MBX 1416 effect in reducing post-prandial insulin and C-peptide peaks will also be evaluated

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be ≥18 to ≤75 years of age at the time of signing the informed consent.
2. Participants must have undergone RYGB or SG surgery at least 12 months prior to study entry.
3. Participants should have a documented history of PBH, defined as Whipple's triad (symptomatic hypoglycemia, capillary glucose ≤54 mg/dL, with symptom resolution by carbohydrate administration) and a minimum of 1 symptomatic hypoglycemic episode per month by patient report.
4. Participants who are either treatment naïve or who are no longer using (i.e., have discontinued as part of their usual medical care) agents known to interfere with glucose metabolism at the time of screening.
5. Participants must have a body mass index (BMI) <45 kg/m2 at screening.
6. Must have signed informed consent.

Exclusion Criteria:

1. History of, or currently active, significant illness or medical disorders that in the opinion of the investigator may preclude participants from participating in the study.
2. Currently on-going type II diabetes mellitus.
3. History of hypoglycemia prior to bariatric surgery.
4. History of insulinoma or other endogenous hyperinsulinemia illness (e.g., congenital hyperinsulinism).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-08-26 (Actual); Primary Completion 2025-12-22 (Estimated); Study Completion 2026-01-26 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline to post-treatment in glucose nadir during a standardized MMTT following different dose levels of MBX 1416. | The duration of the study will be approximately 67 days from screening to end of study (EoS) for any given participant

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - MBX Biosciences Investigational Site, Aurora, Colorado
  - MBX Biosciences Investigational Site, Morehead City, North Carolina
  - MBX Biosciences Investigational Site, Knoxville, Tennessee
  - MBX Biosciences Investigational Site, San Antonio, Texas